CLINICAL TRIAL: NCT06167850
Title: Effect of the Copenhagen Plank on Aductional Strenght and Vertical Jump in Female Football Players: Randomized Controlled Trial
Brief Title: Effect of the Copenhagen Plank on Aductional Strenght and Vertical Jump in Female Football Players
Acronym: ECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina, Clinical Professor, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Clinical trial
Record Dates: First submitted 2023-11-08; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Groin Injury; Muscle Injury
Keywords: Groin pain; Adductors; Copenhagen plank; Strength

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group doing the Copenhagen plank
  Interventions: Procedure: Copenhagen plank
- Control group (No Intervention): Group doesn't do Copenhagen plank

INTERVENTIONS:
Procedure: Copenhagen plank — Performing Copenhagen adduction as prevention for adductor injury.
  Other Names: Copenhagen Adduction
  Arms: Intervention group

SUMMARY:
There is enough evidence to know the high incidence of groin injuries in soccer. Despite this, there is not enough about these in women's football. The researchers perform the Copenhagen plank to obtain an improvement in the improvement of adductor strength and the reduction of groin injuries

DETAILED DESCRIPTION:
At present, there is enough evidence to know the high incidence of groin injuries in soccer. Despite this, there is not enough about them in women's football. Strengthening the adductor muscles is beneficial in preventing these injuries. The Copenhagen plank is beneficial in programs for the prevention and treatment of groin injuries. A randomized controlled trial was carried out. The sample was made up of 26 players between 18 and 31 years of age from the CAP Ciudad de Murcia soccer team. The experimental group (n=12) performed the Copenhagen plank protocol for 4 weeks, the control group continued their training as normal. Performance was assessed using the CMJ jump and the hip adduction strength test using manual dynamometry. 3 measurements were made.

ELIGIBILITY:
Inclusion criteria:

* Girls of legal age
* At least 4.5 hours of weekly training
* Active female soccer team players

Exclusion Criteria:

* Current injury
* Injury in the previous 6 months

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Counter Movement Jump | Up to 12 weeks
  Vertical counter movement jump measured in centimeters
Adductor muscle strength | Up to 12 weeks
  Adductor muscle strength measured in Hz in both legs

CONTACTS AND LOCATIONS:
Locations (1):
- Rocío Martínez Fernández, Murcia, Molina de Segura, Spain

REFERENCES:
- [Background] Walden M, Hagglund M, Ekstrand J. Injuries in Swedish elite football--a prospective study on injury definitions, risk for injury and injury pattern during 2001. Scand J Med Sci Sports. 2005 Apr;15(2):118-25. doi: 10.1111/j.1600-0838.2004.00393.x. PMID 15773867
- [Background] Langhout R, Weir A, Litjes W, Gozeling M, Stubbe JH, Kerkhoffs G, Tak I. Hip and groin injury is the most common non-time-loss injury in female amateur football. Knee Surg Sports Traumatol Arthrosc. 2019 Oct;27(10):3133-3141. doi: 10.1007/s00167-018-4996-1. Epub 2018 Jun 2. PMID 29860603
- [Background] Walden M, Hagglund M, Ekstrand J. UEFA Champions League study: a prospective study of injuries in professional football during the 2001-2002 season. Br J Sports Med. 2005 Aug;39(8):542-6. doi: 10.1136/bjsm.2004.014571. PMID 16046340
- [Background] 4. Harøy J, Clarsen B, Wiger EG, Øyen MG, Serner A, Thorborg K, et al. The Adductor Strengthening Programme prevents groin problems among male football players: a cluster-randomised controlled trial. Br J Sports Med [Internet]. 2019;53(3):150-7. Disponible en: http://dx.doi.org/10.1136/bjsports-2017-098937 5. Jensen J, Hölmich P, Bandholm T, Zebis MK, Andersen LL, Thorborg K. Eccentric strengthening effect of hip-adductor training with elastic bands in soccer players: a randomised controlled trial. Br J Sports Med [Internet]. 2014;48(4):332-8.
- [Background] Watanabe K, Nunome H, Inoue K, Iga T, Akima H. Electromyographic analysis of hip adductor muscles in soccer instep and side-foot kicking. Sports Biomech. 2020 Jun;19(3):295-306. doi: 10.1080/14763141.2018.1499800. Epub 2018 Aug 13. PMID 30102108
- [Background] Ishoi L, Sorensen CN, Kaae NM, Jorgensen LB, Holmich P, Serner A. Large eccentric strength increase using the Copenhagen Adduction exercise in football: A randomized controlled trial. Scand J Med Sci Sports. 2016 Nov;26(11):1334-1342. doi: 10.1111/sms.12585. Epub 2015 Nov 21. PMID 26589483
- [Background] Haroy J, Thorborg K, Serner A, Bjorkheim A, Rolstad LE, Holmich P, Bahr R, Andersen TE. Including the Copenhagen Adduction Exercise in the FIFA 11+ Provides Missing Eccentric Hip Adduction Strength Effect in Male Soccer Players: A Randomized Controlled Trial. Am J Sports Med. 2017 Nov;45(13):3052-3059. doi: 10.1177/0363546517720194. Epub 2017 Aug 14. PMID 28806100
- [Background] Bosco C, Komi PV, Tihanyi J, Fekete G, Apor P. Mechanical power test and fiber composition of human leg extensor muscles. Eur J Appl Physiol Occup Physiol. 1983;51(1):129-35. doi: 10.1007/BF00952545. PMID 6684025
- [Background] Hagglund M, Walden M, Ekstrand J. Injuries among male and female elite football players. Scand J Med Sci Sports. 2009 Dec;19(6):819-27. doi: 10.1111/j.1600-0838.2008.00861.x. Epub 2009 Oct 13. PMID 18980604
- [Background] Holmich P. Long-standing groin pain in sportspeople falls into three primary patterns, a "clinical entity" approach: a prospective study of 207 patients. Br J Sports Med. 2007 Apr;41(4):247-52; discussion 252. doi: 10.1136/bjsm.2006.033373. Epub 2007 Jan 29. PMID 17261557
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Sjovall Anari S, Olsson A, Ohlin A, Desai N, Senorski EH, Sansone M, Lindman I. High-level soccer players have a low rate of return to performance after hip arthroscopy for femoroacetabular impingement syndrome. Knee Surg Sports Traumatol Arthrosc. 2023 Jun;31(6):2071-2078. doi: 10.1007/s00167-023-07336-9. Epub 2023 Mar 22. PMID 36947232
- [Background] 14. Escobar JCZ CCM. Fisioterapia en la pubalgia. Revista de la Federación Española de Medicina del Deporte . 2008;179-88.
- [Background] Holmich P, Larsen K, Krogsgaard K, Gluud C. Exercise program for prevention of groin pain in football players: a cluster-randomized trial. Scand J Med Sci Sports. 2010 Dec;20(6):814-21. doi: 10.1111/j.1600-0838.2009.00998.x. PMID 19883386
- [Background] Collings TJ, Diamond LE, Barrett RS, Timmins RG, Hickey JT, DU Moulin WS, Williams MD, Beerworth KA, Bourne MN. Strength and Biomechanical Risk Factors for Noncontact ACL Injury in Elite Female Footballers: A Prospective Study. Med Sci Sports Exerc. 2022 Aug 1;54(8):1242-1251. doi: 10.1249/MSS.0000000000002908. Epub 2022 Mar 12. PMID 35320148
- [Background] Saad MC, Vasconcelos RA, Mancinelli LVO, Munno MSB, Liporaci RF, Grossi DB. Is hip strengthening the best treatment option for females with patellofemoral pain? A randomized controlled trial of three different types of exercises. Braz J Phys Ther. 2018 Sep-Oct;22(5):408-416. doi: 10.1016/j.bjpt.2018.03.009. Epub 2018 Apr 4. PMID 29661570
- [Background] Thorborg K, Branci S, Nielsen MP, Tang L, Nielsen MB, Holmich P. Eccentric and Isometric Hip Adduction Strength in Male Soccer Players With and Without Adductor-Related Groin Pain: An Assessor-Blinded Comparison. Orthop J Sports Med. 2014 Feb 14;2(2):2325967114521778. doi: 10.1177/2325967114521778. eCollection 2014 Feb. PMID 26535298
- [Background] Yousefzadeh A, Shadmehr A, Olyaei GR, Naseri N, Khazaeipour Z. The Effect of Therapeutic Exercise on Long-Standing Adductor-Related Groin Pain in Athletes: Modified Holmich Protocol. Rehabil Res Pract. 2018 Mar 12;2018:8146819. doi: 10.1155/2018/8146819. eCollection 2018. PMID 29721339
- [Background] 20. Baño Alcaraz A, García Vidal JA, Orcajada Pérez J, Godínez Leal J, Medina i Mirapeix F. Análisis de los desequilibrios musculares de la cadera en corredores aficionados. Eur J Podiatry / Rev Eur Podol [Internet]. 2019;5(2):54-62. Disponible en: http://dx.doi.org/10.17979/ejpod.2019.5.2.5727
- [Background] Krommes K, Petersen J, Nielsen MB, Aagaard P, Holmich P, Thorborg K. Sprint and jump performance in elite male soccer players following a 10-week Nordic Hamstring exercise Protocol: a randomised pilot study. BMC Res Notes. 2017 Dec 4;10(1):669. doi: 10.1186/s13104-017-2986-x. PMID 29202784
- [Background] Kohavi B, Beato M, Laver L, Freitas TT, Chung LH, Dello Iacono A. Effectiveness of Field-Based Resistance Training Protocols on Hip Muscle Strength Among Young Elite Football Players. Clin J Sport Med. 2020 Sep;30(5):470-477. doi: 10.1097/JSM.0000000000000649. PMID 30418198
- [Background] Alonso-Fernandez D, Fernandez-Rodriguez R, Taboada-Iglesias Y, Gutierrez-Sanchez A. Effects of Copenhagen Adduction Exercise on Muscle Architecture and Adductor Flexibility. Int J Environ Res Public Health. 2022 May 27;19(11):6563. doi: 10.3390/ijerph19116563. PMID 35682148
- [Background] Serner A, Jakobsen MD, Andersen LL, Holmich P, Sundstrup E, Thorborg K. EMG evaluation of hip adduction exercises for soccer players: implications for exercise selection in prevention and treatment of groin injuries. Br J Sports Med. 2014 Jul;48(14):1108-14. doi: 10.1136/bjsports-2012-091746. Epub 2013 Mar 19. PMID 23511698